CLINICAL TRIAL: NCT05336279
Title: A Single-center, Single-dose, Randomized, Open-label, Two-cycle, Crossover Study of Bioequivalence of Famitinib Malate Capsules of Different Specifications Taken Orally in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Famitinib Malate in Healthy Volunteers Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-112
Record Dates: First submitted 2022-04-19; First posted 2022-04-20 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: The study is a single-center, single-dose, randomized, open-label, two-cycle, crossover study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group TR (Experimental): T - R
  Interventions: Drug: famitinib malate T(5 mg*4)、famitinib malate R(20 mg)
- Treatment group RT (Experimental): R -T
  Interventions: Drug: famitinib malate T(5 mg*4)、famitinib malate R(20 mg)

INTERVENTIONS:
Drug: famitinib malate T(5 mg*4)、famitinib malate R(20 mg) — TR Group: famitinib malate T on day 1, famitinib malate R on day 13.
  Arms: Treatment group TR
Drug: famitinib malate T(5 mg*4)、famitinib malate R(20 mg) — RT Group: famitinib malate R on day 1, famitinib malate T on day 13.
  Arms: Treatment group RT

SUMMARY:
The study is a single-centre, randomized, open, 2-period, 2-sequence crossover design clinical trial. It is planned to enroll 28 healthy subjects.

Subjects will receive famitinib malate on Day1 and Day13.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects over 18 years old (including the boundary value).
2. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, body mass index (BMI) in the range of 19.0-26.0 kg / m2 (including the critical value).
3. Fertile subjects had no family planning and had to take acceptable contraceptive measures and no plans to donate eggs and sperm within 28 weeks from the date of signing informed consent to the last medication; the serum pregnancy test of fertile women before the enrollment should be negative.
4. The subject can communicate well with the researcher, understand and comply with the requirements of this study, and understand and sign the informed consent.

Exclusion Criteria:

1. Anyone who has suffered from any clinical serious disease such as the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities, or any other disease which can affect the study results.
2. Those who have undergone surgery within 3 months before the trial, or plan to perform surgery during the study period.
3. Those who participate in blood donation within 3 months before screening and donate blood volume ≥ 400 mL or lose blood ≥ 400 mL, participate in blood donation within 1 month before screening and donate blood volume ≥ 200 mL or lose blood ≥ 200 mL, or receive blood transfusion.
4. Have a history of allergies to drugs, food or other substances.
5. Those who have used soft drugs (such as marijuana) within 3 months before screening, or hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before screening; or those with positive results in urine drug abuse screening; or those who have a history of drug abuse or drug dependence within 5 years before screening.
6. Those who have participated in any clinical trials and have taken study drugs within 3 months before the first administration.
7. Those who have taken any medicine within 4 weeks before the first administration (including prescription medicines, non-prescription medicines, Chinese herbal medicines, vitamins, calcium tablets and other food supplements).
8. Those who smoke more than 5 cigarettes per day within 3 months before screening and could not stop using any tobacco products during the trial.
9. Regular drinkers within 6 months before screening, that is, drinking more than 14 g of alcohol per week (1 g alcohol ≈ 360 mL of beer, or 45 mL of spirits with 40% alcohol content, or 150 mL of wine), and any alcohol-containing products cannot be stopped during the study, and those with positive results in alcohol breath test.
10. Vital signs, vital signs, physical examination, 12-lead electrocardiogram, chest X-ray, abdominal ultrasound and clinical laboratory tests with abnormalities and clinical significance.
11. HBsAg positive, HCVAb positive, HIV antibody positive, syphilis antibody positive.
12. 48 hours before the first dose until the end of the study, those who refuse to stop any beverages or foods containing methylxanthines, such as coffee, tea, cola, chocolate, etc.; 7 days before the first dose until the end of the study, those who refuse to stop using any beverage or food containing grapefruit; has special dietary requirements and cannot comply with the unified diet.
13. Those who have been vaccinated against 2019-nCOV, other inactivated or attenuated vaccines within 28 days before the first administration, or who plan to be vaccinated against 2019-nCoV during research.
14. Those with a history of fainting of blood or needles and intolerance to venipuncture.
15. Lactating women.
16. The researchers considered that the subjects had any other factors that were not suitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Famitinib | from Day1 to Day9 after the first cycle （each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Area under the plasma concentration versus time curve (AUC0-t) of Famitinib | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Area under the plasma concentration versus time curve (AUC0-∞) of Famitinib | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) of Famitinib | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Elimination half-life (T1/2) of Famitinib | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Apparent oral clearance (CL/F) of Famitinib | from Day1 to Day9（each cycle is 9 days） after the first cycle and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Maximum observed plasma concentration (Cmax) of SHR116637 | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Area under the plasma concentration versus time curve (AUC0-t) of SHR116637 | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Area under the plasma concentration versus time curve (AUC0-∞) of SHR116637 | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Time to maximum observed plasma concentration (Tmax) of SHR116637 | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Time to elimination half-life (T1/2) of SHR116637 | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Apparent oral clearance (CL/F) of SHR116637 | from Day1 to Day9 after the first cycle（each cycle is 9 days） and from Day13 to Day21 after the second cycle（each cycle is 9 days）
Number of subjects with adverse events and the severity of adverse events | from Day1 to Day21 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of USTC, Jinan, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided